CLINICAL TRIAL: NCT00809913
Title: Relevance of Biomarkers and Clinical Predictors of Outcome in Unselected Population With Febrile Urinary Tract Infection at Primary Care and Emergency Department in a Prospective, Randomized Cohort Trial Comparing Short (7 Days) Antibiotic Treatment With Conventional Treatment (14 Days)
Brief Title: Febrile Urinary Tract Infection Randomized Short Treatment Trial
Acronym: FUTIRST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Bronovo Hospital (Other); Medical Center Haaglanden (Other); Spaarne Gasthuis (Other); Rijnland Hospital (Other); Diaconessenhuis Leiden (Unknown); Groene Hart Ziekenhuis (Other)
Responsible Party: Principal Investigator, C. van Nieuwkoop, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL22172.058.08
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Tract Infection
Keywords: Urinary Tract Infection; Fever; Acute Pyelonephritis; Treatment duration; Febrile Urinary Tract Infection Treatment Duration
MeSH Terms: conditions — Urinary Tract Infections; Fever | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short treatment (Experimental): 7 days of standard antibiotic treatment (preferably ciprofloxacin) followed by 7 days of placebo
  Interventions: Drug: short treatment (ciprofloxacin)
- Standard treatment (Active Comparator): 14 days of standard antibiotic treatment (initial b-lactam or fluoroquinolone followed by ciprofloxacin through the 8th till 14th day)
  Interventions: Drug: short treatment (ciprofloxacin)

INTERVENTIONS:
Drug: short treatment (ciprofloxacin) — 7 days of antibiotic treatment for febrile urinary tract infection / acute pyelonephritis compared to standard treatment of 14 days

SUMMARY:
The purpose of this study is to determine whether a 7-day duration of antibiotic treatment of febrile urinary tract infection (FUTI) is non inferior to 14-day standard duration of treatment in unselected population presenting at primary care or emergency department.

DETAILED DESCRIPTION:
In the last decades hospitalization rates of patients with acute pyelonephritis (AP) or FUTI has decreased from almost 100% to 10-30%. The outpatient management of patients with FUTI has become popular as well as oral antimicrobial treatment regiments and shortening of treatment duration. However, as such approaches are only discovered in otherwise young health non-pregnant women, the best management of FUTI in the elderly, men and patients with co-morbidity remains elusive. Bases on personal perception of the attending physician antibiotic treatment, duration varies approximately between 7-14 days. Facing the aging of the general population, it is urgent to better define the optimal treatment for AP or FUTI in an unselected population and to identify those at risk for treatment failure or poor outcome to guide and optimize individual patient management and to prevent on the one hand unnecessary long treatment duration and hospital admission and on the other hand unsafe short duration or unsafe outpatient management.

In this study the efficacy and safety of a 7-day antimicrobial regimen compared to a 14-day antimicrobial regimen will be evaluated in an unselected population presenting with FUTI at primary care or emergency department. In addition a clinical and/or biomarker based scoring system of disease severity will be derived to predict those at risk for treatment failure or poor outcome.

ELIGIBILITY:
Inclusion Criteria:

* Competent patient aged 18 years or above
* One or more symptom(s) suggestive of urinary tract infection (dysuria, frequency or urgency*; perineal or suprapubic pain; costo-vertebral tenderness or flank pain)
* Fever (ear or rectal temp of 38.2 oC or higher, or axillary temp of 38 oC or higher), or history of feeling feverish with shivering or rigors in the past 24 hours
* Positive urine nitrate test and/or leucocyturia as depicted by positive leukocyte esterase test or microscopy

Exclusion Criteria:

* Known allergy to fluoroquinolones
* Female patients who are pregnant or lactating
* Patients with known polycystic kidney disease
* Patients on permanent renal replacement therapy (hemodialysis or peritoneal dialysis)
* Patients with history of kidney transplantation
* Residence outside country of enrolment
* Inability to speak or read Dutch
* Isolated causal uropathogen resistant to ciprofloxacin
* Renal abscess
* Chronic bacterial prostatitis
* Suspicion or evidence of any metastatic infectious foci

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-12; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate through the 10- to 18-day posttherapy visit. Clinical cure is defined as the resolution of fever and signs and symptoms of UTI. | 10-18 day posttherapy

SECONDARY OUTCOMES:
Microbiological cure rate 10- to 18-day posttherapy | 10-18 day posttherapy
All cause mortality | 30 and 90 days
Clinical cure rate 70- to 84- day posttherapy | 70-84 days posttherapy
Relapse rate of any urinary tract infection | 90 days
Adverse events | 90 days
Rate of pelvic floor dysfunction as assessed by standardized questionaire | 10-18 days posttherapy
Occurence of Clostridium Difficile associated diarrhea | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jaap T. van Dissel, MD, PhD, Study Chair — Leiden University Medical Center; Cees van Nieuwkoop, MD, PhD, Principal Investigator — Leiden University Medical Center and Haga Hospital
Locations (6):
- Netherlands (6):
  - Groene Hart Hospital, Gouda
  - Leiden University Medical Center, Leiden
  - Alrijne Hospital, Leiden
  - Alrijne Hospital, Leiderdorp
  - Medical Center Haaglanden, The Hague
  - Bronovo Hospital, The Hague

REFERENCES:
- [Background] van Nieuwkoop C, van't Wout JW, Assendelft WJ, Elzevier HW, Leyten EM, Koster T, Wattel-Louis GH, Delfos NM, Ablij HC, Kuijper EJ, Pander J, Blom JW, Spelt IC, van Dissel JT. Treatment duration of febrile urinary tract infection (FUTIRST trial): a randomized placebo-controlled multicenter trial comparing short (7 days) antibiotic treatment with conventional treatment (14 days). BMC Infect Dis. 2009 Aug 19;9:131. doi: 10.1186/1471-2334-9-131. PMID 19691829
- [Derived] Stalenhoef JE, van Nieuwkoop C, Wilson DC, van der Starre WE, van der Reijden TJK, Delfos NM, Leyten EMS, Koster T, Ablij HC, van 't Wout JJW, van Dissel JT. Procalcitonin, mid-regional proadrenomedullin and C-reactive protein in predicting treatment outcome in community-acquired febrile urinary tract infection. BMC Infect Dis. 2019 Feb 14;19(1):161. doi: 10.1186/s12879-019-3789-6. PMID 30764769
- [Derived] van Nieuwkoop C, van der Starre WE, Stalenhoef JE, van Aartrijk AM, van der Reijden TJ, Vollaard AM, Delfos NM, van 't Wout JW, Blom JW, Spelt IC, Leyten EM, Koster T, Ablij HC, van der Beek MT, Knol MJ, van Dissel JT. Treatment duration of febrile urinary tract infection: a pragmatic randomized, double-blind, placebo-controlled non-inferiority trial in men and women. BMC Med. 2017 Apr 3;15(1):70. doi: 10.1186/s12916-017-0835-3. PMID 28366170